CLINICAL TRIAL: NCT00294814
Title: Gas and Solid Brain Microembolization Detected by the EmbodopR TCD System During Proximal Coronary Graft Anastomosis Done With Aortic Cross Clamping, Partial Occlusion or the HeartstringR Device and Their Effect on Neurocognitive Performance After Coronary Bypass Operation
Brief Title: TCD Detection of Gas and Solid Micro-Emboli in Patients Undergoing Coronary Artery Bypass Grafting (CABG): The Influence of Proximal Anastomosis Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMBO_CTIL
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2006-05

CONDITIONS: Intracranial Embolism and Thrombosis; Postoperative Complications
Keywords: Cardiac Surgery; CABG; Microemboli; Transcranial Doppler; Cognitive Decline; Anastomotic Device; Proximal Anastomosis; Coronary Artery Bypass Graft (CABG)
MeSH Terms: conditions — Intracranial Embolism and Thrombosis; Postoperative Complications; Cognitive Dysfunction

INTERVENTIONS:
Device: Proximal anastomosis using Heartstring anastomotic device

SUMMARY:
The purpose of this study is to test the hypothesis that using three different techniques to anastomose coronary grafts to the aorta: partial occlusion, single cross clamp, or using the Heartstring anastomotic device, will change the amount of gas and solid microemboli as detected by the EmbodopR transcranial Doppler (TCD) system and consequently the neurocognitive performance of patients after coronary bypass operation.

DETAILED DESCRIPTION:
It is not uncommon for a cardiac surgical patient to have his heart fixed but his brain damaged. Sometimes the damage is overt and manifests itself as a major neurological deficiency. The frequency of stroke, the so called type 1 damage, is reported to be between 1 and 4 percent. This may increase mortality from 1.4% to 22% and hospitalization from 6.6 days to 17.5 days. Diffuse encephalopathy, presenting as delirium, confusion, coma and seizures, so called type 2 damage, is reported to appear in a much higher frequency of 3% to 7%, depending on timing and methods of evaluation. This type of damage will increase mortality from 1.4% to 7.5% and hospitalization from 6.6% to 15.2%. Sometimes it is more subtle and appears as neurocognitive decline. This type of damage may be found in 53% of the patients at discharge, in 24% after six months and the frequency rises again to 42% at five years. The impact on the patient and his family might be devastating and the burden on the medical system and society enormous. Long term, moderate to severe disability may affect 69% of the stroke patients and survival may decline to 67% after one year.

After years of research efforts it became evident that inadequate global blood flow to the brain is relatively uncommon and cerebral hemorrhage is a rare cause of brain damage during cardiac operations. It also became evident that one of the most important damage mechanisms is embolization to the brain and the inflammatory response which amplifies the ischemic embolic damage. Looking for possible embolic sources by monitoring embolic signals (HITS) on the transcranial doppler (TCD) tracings, researchers found that manipulation of the aorta during cardiac surgery, like cannulation and especially clamping is a major source of emboli. Using the side biting clamp while performing proximal anastomosis has the potential to crush the aortic wall and release macro and micro emboli especially when the aorta is atherosclerotic. Using a single cross clamp technique might eliminate the aortic wall solid debris but introduce air emboli instead.

Dealing with the same problem, a few proximal anastomotic devices have been introduced and most of them withdrawn from the market because of inferior patency rate. The Heartstring proximal anastomotic device is one of the recently introduced devices for which early good patency rate has been demonstrated. The advantages, in terms of less brain embolization or improved neurologic outcome, have never been demonstrated for the Heartstring or any other anastomotic device.

A recent potential breakthrough in this field of emboli research and prevention in order to improve neurologic outcome after cardiac surgery is the introduction of the EmbodopR system by DWL. This is a high quality TCD system which has been further developed to monitor cerebral emboli. It contains a module which automatically screens every event suspected as embolic, eliminates those recognized as artifacts according to four different criteria and records only real embolic events. Another module can differentiate every event as gas or solid emboli by simultaneously insonating the middle cerebral artery blood with tow ultrasound beams, each of different frequency. The result is a new ability for real time monitoring and characterization of embolic events during cardiac operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for surgical coronary revascularization at the Department of Cardiac Surgery of Rambam Medical Center, Haifa, Israel.
* Patients should be conscious and cooperative to perform neurocognitive evaluation.

Exclusion Criteria:

* Patients that lack "temporal window" for TCD monitoring will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100

PRIMARY OUTCOMES:
Number of gas\solid microemboli detected by TCD
Neurocognitive performance

SECONDARY OUTCOMES:
Mortality
Organ failure (including brain damage)
Intensive care unit (ICU) length of stay\hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Adler, MD, Study Director — Rappaport Faculty of Medicine; Simcha Milo, Prof., Study Chair — Rappaport Faculty of Medicine; Majed Kabaha, MD, Principal Investigator — Cardiac Surgery Dep. Rambam Medical Center
Locations (1):
- Dr Zvi Adler, Haifa, Israel